CLINICAL TRIAL: NCT01252381
Title: The Importance of Supplementary Intake of Vitamin D on the Efficacy of 12 Weeks of Strength Training in Both Vitamin D Sufficient Younger and Older People
Brief Title: Supplementary Intake of Vitamin D During 12 Weeks Strength Training in Younger and Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Institute of Sports Medicine, Copenhagen (Unknown)
Responsible Party: Principal Investigator, Jakob Agergaard, MSc, PhD Student, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BBH 77
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Muscle Strength; Tendon Elasticity; Muscle CSA; Tendon CSA; VDR Receptor

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vitamin D (Active Comparator)
  Interventions: Other: 12 weeks Strength exercise training
- Calcium tablet (Placebo Comparator)
  Interventions: Other: 12 weeks Strength exercise training

INTERVENTIONS:
Other: 12 weeks Strength exercise training — Training 3 times a week, leg extensions and leg press

SUMMARY:
The aim is to investigate the importance of vitamin D levels to achieve the effect of strength training. If we can show that vitamin D has an effect of training, the ultimate goal is to find out why and how vitamin D affects muscle.

This would potentially have important implications for public health. Since a large number of populations, including elderly, are shown to have too little vitamin D and also has low muscle strength, it will be essential that these people added vitamin D in relation to training and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Men 20-30 or 60-75 years old

Exclusion Criteria:

* smokers Knee problems On medication affecting protein synthesis High exposure to sun light (ex. ski holiday) during the trial

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area of thigh musculature and knee tendon | 12 weeks
VDR potential target CYP27b1 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine - Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Agergaard J, Trostrup J, Uth J, Iversen JV, Boesen A, Andersen JL, Schjerling P, Langberg H. Does vitamin-D intake during resistance training improve the skeletal muscle hypertrophic and strength response in young and elderly men? - a randomized controlled trial. Nutr Metab (Lond). 2015 Sep 30;12:32. doi: 10.1186/s12986-015-0029-y. eCollection 2015. PMID 26430465